CLINICAL TRIAL: NCT01814930
Title: Evaluation of a Brief Standardized Postpartum Counseling Intervention's Effect on Repeat Pregnancy Rates Contraceptive Choice/Use/Continuation/Satisfaction in Adolescents
Brief Title: Adolescent Postpartum Contraceptive Counseling Intervention
Acronym: PPCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Courtney Schreiber, Director, Fellowship in Family Planning, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 814909
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Adolescent Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Care (No Intervention): Routine postpartum contraceptive counseling
- Individual counseling (Experimental): Brief standardized contraceptive counseling intervention
  Interventions: Behavioral: Brief standardized contraceptive counseling intervention

INTERVENTIONS:
Behavioral: Brief standardized contraceptive counseling intervention — The intervention employed an in-person counseling strategy that included empowerment messaging and an instrument to clarify the participants' preferences for contraception in the context of their goals for future childbearing.
  Arms: Individual counseling

SUMMARY:
Postpartum contraceptive counseling varies widely in its provision; no standardized practice has been well-established by the literature. We intend to evaluate how directed postpartum contraceptive counseling to adolescents aged 14-19 affects key outcomes over time. Subjects will be randomized to receive either the standardized contraceptive counseling intervention or routine postpartum care. We will then assess the difference in repeat pregnancy rates between the two groups

ELIGIBILITY:
Inclusion Criteria:

* 14-19 years old
* primiparous
* immediately postpartum
* delivery of a full term live singleton infant (>37 weeks) at HUP

Exclusion Criteria:

* not planning to reside in/near Philadelphia for the next year

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is repeat pregnancy rate | 1 year
  Repeat pregnancy rate of intervention and control groups will be assessed

SECONDARY OUTCOMES:
Contraceptive choice, use and continuation rates postpartum as well as contraceptive satisfaction rates | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Courtney A Schreiber, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Frarey A, Gurney EP, Sober S, Whittaker PG, Schreiber CA. Postpartum contraceptive counseling for first-time adolescent mothers: a randomized controlled trial. Arch Gynecol Obstet. 2019 Feb;299(2):361-369. doi: 10.1007/s00404-018-4969-0. Epub 2018 Nov 23. PMID 30470924